CLINICAL TRIAL: NCT04684615
Title: Mental Health Impact of the COVID-19 Pandemic on Amish and Mennonite Participants in AMBiGen
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000038; 000038-M
Record Dates: First submitted 2020-12-23; First posted 2020-12-24 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05-15

CONDITIONS: Depression; Anxiety; Bipolar Disorder
Keywords: Anabaptist; Coronavirus; behavioral health; Mood Disorder; Natural History
MeSH Terms: conditions — Depression; Anxiety Disorders; Bipolar Disorder; Coronavirus Infections; Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AmBiGen: Individuals who are enrolled in AmBiGen over the last 3 years

SUMMARY:
People have had to make a lot of changes to their lives due to the COVID-19 health crisis. Most experts agree that social distancing and other safety measures have taken a toll on people s mental health. Amish and Mennonite communities often have large families. They may have limited access to health care. Their lifestyle is based on interaction and group events rather than technology. So people in Amish and Mennonite communities may experience the pandemic in their own special ways.

Objective:

To describe the relationship between stress related to the pandemic and self-rated measures of mental health symptoms and distress among Amish and Mennonite people with bipolar disorder and related conditions, and their family members.

Eligibility:

Adults ages 18 and older who are taking part in the NIMH AMBiGen study (80-M-0083).

Design:

Participants will be mailed 4 surveys. One survey will ask about depression symptoms. One survey will ask about mania symptoms. One survey will assess a broad range of psychological problems. One survey will assess the impact of COVID-19 on their mental health. They will fill out the surveys 4 times over 24 months.

The surveys will not include participants names, just codes. This will help protect privacy.

Data collected in 80-M-0083 will be used. This includes data about participants genes, medical conditions, and assessments.

Participants will get an 800 number they can call to speak to the research team. They can also write to the team if they prefer. Participants who wish will get referrals for mental health services. Participation will last up to 24 months. There will be an option for recontact in the future.

DETAILED DESCRIPTION:
This protocol leverages existing NIMH studies and participants to accomplish time-sensitive research on the mental health impact of environmental stressors imposed by the COVID-19 pandemic. The study will describe the relationship between stressors related to COVID-19 and self-rated measures of mental health symptoms and distress among Amish and Mennonite participants in an ongoing study of bipolar disorder (AMBiGen), and their family members.

Objectives: The primary objective is to describe the relationship between stressors related to COVID-19 and self-rated measures of mental health symptoms and distress among individuals with bipolar disorder, related conditions, and their family members. The secondary objectives are to determine the roles played by psychiatric diagnosis, genetic risk of various mental illnesses, and perceived social support in moderating risk and resilience for mental health during and after the COVID-19 pandemic.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Active enrollment in Protocol 80-M-0083
2. 18 years of age and older.

EXCLUSION CRITERIA:

1. Under age 18.

INCLUSION OF VULNERABLE PARTICIPANTS:

The study will be not be targeting any vulnerable populations. We are not planning to recruit children; all participants being invited to participate have previously been assessed under Protocol 80-M-0083 as over the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample size will be up to 1,000 and will include participants 18 years and older of both sexes, any gender, and health status. This sample size is an estimate of the number of individuals who have enrolled the NIMH AmBiGen study in the past and might respond if re-contacted, as well as family members who may not have enrolled in the past but are expected to share genetic, familial, and community risk/resilience factors.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
To describe the relationship between stressors related to COVID-19 and self-rated measures of mental health symptoms and distress among a range of participants including various patient populations and healthy volunteers. | assesses the stressors experienced as a result of the COVID-19 pandemic.
  The availability of repeated measurement will allow us to establish whether changes in stressors related to COVID-19 are associated with changes in mental health symptoms and distress within subject.

SECONDARY OUTCOMES:
1) Determine whether existing mental health concerns moderates the relationship between stressors related to COVID-19 and self-rated measures of mental health symptoms and distress. 2) To identify risk and resilience factors among study particip... | End of study
  In order to determine whether the participant has existing mental health concerns, we must collect information on a variety of symptoms related to mental health. We hypothesize that certain participant- level characteristics may be related to the mental health and behavioral impacts of the COVID-19 pandemic. For this exploratory aim, we will evaluate a variety of sociodemographic, clinical, genetic, and behavioral variables.

CONTACTS AND LOCATIONS:
Overall Officials: Francis J McMahon, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States